CLINICAL TRIAL: NCT04254198
Title: Tertulias: Addressing Social Isolation to Reduce Depression Among Women of Mexican Origin
Brief Title: Tertulias Social Isolation Women's Groups Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Janet M Page-Reeves, Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-160; 1R01MD014153-01 (NIH)
Record Dates: First submitted 2019-09-26; First posted 2020-02-05 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Social Isolation; Depression
Keywords: Immigrant; Women; Peer support group; Community-engaged
MeSH Terms: conditions — Social Isolation; Depression

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Modified Attention Placebo Control
  Interventions: Behavioral: Modified Attention Placebo Control (MAPC)
- TERTULIAS structured dialogue peer support groups (Experimental): Structured Dialogue peer support group
  Interventions: Behavioral: TERTULIAS structured dialogue peer support groups

INTERVENTIONS:
Behavioral: TERTULIAS structured dialogue peer support groups — TERTULIAS will involve structured dialogue groups using the model developed and tested by the investigators through their preliminary research. Each group will have 10 women and will meet weekly for two hours over a 12-month period. Group meetings will be conducted in Spanish, led by a team of two FMI facilitators. Facilitation will use the structured dialogue approach. In the last two months of each cohort, participants will be invited to write their own stories or recipes, or produce poetry or art representing their experience to share with the group. These contributions will be gathered and reproduced in "booklet" form and each participant will receive a copy.
  Arms: TERTULIAS structured dialogue peer support groups
Behavioral: Modified Attention Placebo Control (MAPC) — MAPC participants will receive a phone call every other month from the project coordinator to document that their contact information is up to date, to remind them that they are in the study and to tell them that the study is continuing. Survey data and hair samples will be gathered from them at baseline and 12 months
  Arms: Control

SUMMARY:
This study will use a multi-level, community-engaged approach to implement "TERTULIAS" ("conversational gatherings" in Spanish). The intervention uses an innovative, culturally and contextually situated peer support group design that was developed by the investigators to improve health outcomes and reduce health disparities for female mexican immigrant (FMI) participants in Albuquerque, New Mexico. The study will use a rigorous, transdisciplinary, QUAL⇒QUANT, mixed-method research design. The investigators will document results of the intervention on the primary hypotheses of a decrease in depression, and increases in resilience and social support, as well as on the secondary hypotheses of decreased stress (including the use of innovative testing of hair cortisol as a biomarker for chronic stress), and an increase in social connectedness and positive assessment of knowledge and empowerment gained through the TERTULIAS intervention.

DETAILED DESCRIPTION:
Specific Aims. The investigators will conduct a randomized controlled trial with 240 FMIs. Intervention participants will attend a weekly peer group session over 12 months. Control group participants will receive a bimonthly check-in call. All will be surveyed using validated instruments and give hair samples gathered at baseline and 12 months. A subset will be interviewed, and group sessions will be documented. Data will be triangulated using different methods with a QUAL⇒QUAN simultaneous data collection and analysis approach to integrate, converge, and elaborate findings in a way that would not be feasible using only one method.

Aim 1. To measure whether a culturally situated peer group intervention will reduce depression and stress associated with the experience of immigration. Question: Does an intervention design that reproduces culturally important interactions, activities, and constructs lost through immigration result in decreased participant depression and stress? Hypothesis: Incorporating peer-to-peer social interaction, food sharing, and storytelling into the design of a nonclinical peer support group intervention will leverage positive aspects of participant culture and create an experiential context that will (a) decrease participant depression scores by at least 6.5 points more on the Center for Epidemiologic Studies Depression Scale (CES-D) as compared to controls (effect size Cohen's d = 0.43), and (b) lower stress scores in participants more than in controls with d ≥ 0.5 as measured by the Perceived Stress Scale (PSS). The investigators will also assess stress using a cutting-edge biological assessment of hair cortisol as a biomarker for chronic stress.

Aim 2. To test whether an intervention using a "women's funds of knowledge" approach results in improved resilience, knowledge and empowerment. Question: Does an intervention design that encourages participants to share knowledge they developed through life experience and that values this knowledge as a form of expertise nurture protective factors (resilience and knowledge/empowerment) to help FMIs adapt to the immigration context and disrupt the mechanisms that produce health disparities? Hypothesis: Incorporating, valuing and validating women's knowledge and experience in the design of a peer support group intervention will improve participant capacity to adapt to the immigrant context and provide participants with empowering knowledge to deal with new situations. Intervention participants will have higher scores at 12 months and have a larger increase over time as compared to controls (d = 0.5) on the Connor-Davidson Resilience Scale-25 ("CD-RISC 25"). Knowledge and empowerment will be assessed at 12 months and expect to find high scores with the Trauma-Informed Practice (TIP) Scale (which is designed for post-use).

Aim 3. To investigate whether a culturally situated peer group intervention using a women's funds of knowledge approach can give participants' a sense and experience of social and physical connection ("emplacement") that is lost in the process of immigration. Question: Can the proposed peer support group intervention recreate social and physical connections lost through immigration and strengthen participant social networks? Hypothesis: The peer group will create a culturally appropriate context for establishing interpersonal connections between group members and will give participants a sense of belonging within a social and contextual milieu. At study end, (a) experimental participants will have a marked increase in social support scores v.s. the control group using the Medical Outcomes Study Social Support Survey (MOS SSS) (d ≥ 0.5), and (b) stronger, more dense social connections as described by a social network analysis.

Project Outcomes. This intervention with FMIs will test an innovative intervention to reduce social isolation as a mechanism for reducing depression by leveraging positive cultural dynamics and women's funds of knowledge to nurture social connectedness, knowledge, and resiliency factors in the lives of participants in a transformative way. Generalizability. This trial of TERTULIAS will create a replicable, scalable model for culturally appropriate health promotion with FMIs that has implications for health promotion work with other women from recent and first generation immigrant populations.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* Female immigrant
* Born in Mexico
* Reports household income under 250% Federal Poverty Level
* Speaks Spanish fluently

Exclusion Criteria:

* prisoners
* individuals unable to consent
* children

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 241 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Page-Reeves, PhD, Principal Investigator — UNM Dept. of Family and Community Medicine
Locations (2):
- United States (2):
  - Centro Savila, Albuquerque, New Mexico
  - One Hope Centro De Vida Health Center, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Page-Reeves J, Murray-Krezan C, Regino L, Perez J, Bleecker M, Perez D, Wagner B, Tigert S, Bearer EL, Willging CE. A randomized control trial to test a peer support group approach for reducing social isolation and depression among female Mexican immigrants. BMC Public Health. 2021 Jan 11;21(1):119. doi: 10.1186/s12889-020-09867-z. PMID 33430845

RESULTS

PARTICIPANT FLOW:
Groups:
- TERTULIAS structured dialogue peer support groups: Structured Dialogue peer support group
  Tertulias structured dialogue peer support groups: TERTULIAS will involve structured dialogue groups using the model developed and tested by the investigators through their preliminary research. Each group will have 10 women and will meet weekly for two hours over a 12-month period. Group meetings will be conducted in Spanish, led by a team of two females of Mexican origin facilitators. Facilitation will use the structured dialogue approach. In the last two months of each cohort, participants will be invited to write their own stories or recipes, or produce poetry or art representing their experience to share with the group. These contributions will be gathered and reproduced in "booklet" form and each participant will receive a copy.
Period: Overall Study
Arm/Group | Control | TERTULIAS structured dialogue peer support groups
Started | 117 | 124
Completed | 111 | 106
Not Completed | 6 | 18

BASELINE CHARACTERISTICS:
Population: The Intention-to-Treat (ITT) population is all participants who were randomized and completed the baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | TERTULIAS Structured Dialogue Peer Support Groups | Total
Number analyzed (Participants) | 117 | 124 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (10.9) | 47.6 (10.6) | 48.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 124 | 241
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 117 | 124 | 241
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 117 | 124 | 241
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 117 | 124 | 241
Marital Status [Count of Participants; unit: Participants]
  Married/partnered | 75 | 64 | 139
  Single/divorced/separated/widowed | 42 | 60 | 102
Number of children [Mean (Standard Deviation); unit: children] | 2.7 (1.3) | 2.7 (1.4) | 2.7 (1.3)
Family or friends living in same location [Count of Participants; unit: Participants] | 113 | 120 | 233
Speaks english [Count of Participants; unit: Participants] | 52 | 66 | 118
Employed [Count of Participants; unit: Participants] | 67 | 77 | 144
Overall Health Status [Count of Participants; unit: Participants]
  Well | 81 | 89 | 170
  Not well | 36 | 35 | 71
Depression score (CES-D) [Mean (Standard Deviation); unit: units on a scale] — Summed scores of the 20-item Center for Epidemiologic Studies Depression Scale (CES-D). Summed scores range from 0 to 100 with higher scores indicating higher levels of depression.
  units on a scale | 16.0 (11.9) | 16.4 (12.0) | 16.2 (11.9)
Resilience (CD-RISC) [Mean (Standard Deviation); unit: units on a scale] — Summed scores of the 25-item Connor-Davidson Resilience Scale-25 (CD-RISC 25).Summed scores range from 0 to 100 with higher scores indicating higher levels of resilience.
  units on a scale | 82.4 (14.1) | 80.6 (14.6) | 81.5 (14.3)
Social Support (MOS-SS) [Mean (Standard Deviation); unit: units on a scale] — Total scaled scores of the 19-item Medical Outcomes Study Social Support Survey (MOS SSS).Total scaled scores range from 0 to 100 with higher scores indicating higher levels of social support
  units on a scale | 83.7 (15.3) | 80.3 (17.7) | 81.9 (16.6)
Perceived Stress (PSS-14) [Mean (Standard Deviation); unit: units on a scale] — Summed scores of the 14-item Perceived Stress Scale (PSS-14). Summed scores range from 0 to 56 with higher scores indicating higher levels of stress.
  units on a scale | 33.9 (6.6) | 34.4 (6.5) | 34.2 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression
Description: Comparison of intervention and control participants of their change in depression scores between baseline and 12 months as measured by the summed scores of the 20-item Center for Epidemiologic Studies Depression Scale (CES-D). Summed scores range from 0 to 100 with higher scores indicating higher levels of depression. Changes will be measured as 12 months - Baseline, so negative change scores indicate decreased depression.
Time Frame: Baseline, 12 months
Population: From the Intention-to-Treat (ITT) population, all participants who were randomized and completed the baseline assessment, and who also completed the 12-month follow-up assessment.
Measure: Least Squares Mean (98.3% Confidence Interval); unit: units on a scale
Arm/Group | Control | TERTULIAS structured dialogue peer support groups
Number analyzed (Participants) | 111 | 106
units on a scale | -2.01 [-4.70 to 0.69] | -5.10 [-7.85 to -2.35]
Statistical Analysis 1: Comparison: Control vs TERTULIAS structured dialogue peer support groups; Test type: Superiority; p = 0.0473, Mixed Models Analysis — To adjust for multiplicity due to three primary outcomes, the p-value should be compared to a Bonferroni-corrected type-I error level of 0.05/3 = 0.017; Model is adjusted for cohort, site, marital status, and overall health status; Slope = 0.231, 98.3% CI 2-sided [-0.0474 to 0.509], Standard Error of Mean 0.116 — The beta coefficient (0.231) is for the treatment x time interaction effect on log-transformed CES-D scores. Delta method used for calculating confidence intervals for the Least Squares (LS) Mean changes over time per arm with cov=compound symmetry

2. Primary Outcome: Change in Resilience
Description: Comparison of intervention and control participants of their change in resilience scores between baseline and 12 months as measured by the summed scores of the 25-item Connor-Davidson Resilience Scale-25 (CD-RISC 25).Summed scores range from 0 to 100 with higher scores indicating higher levels of resilience. Changes will be measured as 12 months - Baseline, so positive change scores indicate increased resilience.
Time Frame: Baseline, 12 months
Population: as for outcome 1
Measure: Least Squares Mean (98.3% Confidence Interval); unit: units on a scale
Arm/Group | Control | TERTULIAS structured dialogue peer support groups
Number analyzed (Participants) | 111 | 106
units on a scale | -0.27 [-3.68 to 3.15] | 5.08 [1.68 to 8.48]
Statistical Analysis 1: Comparison: Control vs TERTULIAS structured dialogue peer support groups; Test type: Superiority; p = 0.0067, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Model is adjusted for cohort, site, overall health status and the interaction between cohort and site; Slope = 0.383, 98.3% CI 2-sided [0.0464 to 0.720], Standard Error of Mean 0.140 — The beta coefficient (0.383) is for the treatment x time interaction effect on log-transformed CD-RISC scores. Delta method used for calculating confidence intervals for the LS Mean changes over time per arm with cov=compound symmetry

3. Primary Outcome: Change in Social Support
Description: Comparison of intervention and control participants of their change in social support scores between baseline and 12 months as measured by the total scaled scores of the 19-item Medical Outcomes Study Social Support Survey (MOS SSS).Total scaled scores range from 0 to 100 with higher scores indicating higher levels of social support. Changes will be measured as 12 months - Baseline, so positive change scores indicated increased social support.
Time Frame: Baseline, 12 months
Population: as for outcome 1
Measure: Least Squares Mean (98.3% Confidence Interval); unit: units on a scale
Arm/Group | Control | TERTULIAS structured dialogue peer support groups
Number analyzed (Participants) | 111 | 106
units on a scale | 0.45 [-3.47 to 4.37] | 6.56 [2.34 to 10.77]
Statistical Analysis 1: Comparison: Control vs TERTULIAS structured dialogue peer support groups; Test type: Superiority; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Generalized linear mixed model with beta distribution, adjusted for cohort, site, overall health status and interaction between arm and cohort; Slope = -0.747, 98.3% CI 2-sided [-1.215 to -0.280], Standard Error of Mean 0.194 — The beta coefficient (-0.747) is for the treatment x time interaction effect on MOS-SS scores on a logit scale. The CIs for the LS Mean changes over time per arm were estimated via the delta method and are reported on the original MOS-SS scale

4. Secondary Outcome: Change in Perceived Stress
Description: Comparison of intervention and control participants of their change in social support scores between baseline and 12 months as measured by the summed scores of the 14-item Perceived Stress Scale (PSS-14). Summed scores range from 0 to 56 with higher scores indicating higher levels of stress. Changes will be measured as 12 months - Baseline, so negative change scores indicate decreased perceived stress.
Time Frame: Baseline, 12 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Control | TERTULIAS structured dialogue peer support groups
Number analyzed (Participants) | 111 | 106
units on a scale | -1.36 [-3.04 to 0.33] | -0.44 [-2.13 to 1.24]
Statistical Analysis 1: Comparison: Control vs TERTULIAS structured dialogue peer support groups; Test type: Superiority; p = 0.4510, Mixed Models Analysis — P-value not adjusted for multiple comparisons; Model is adjusted for cohort and site; Slope = -0.913, 95% CI 2-sided [-3.82 to 2.00], Standard Error of Mean 1.21 — The beta coefficient (-0.913) is for the treatment x time interaction effect on non-transformed PSS scores

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse events were documented.
Arm/Group | Control | TERTULIAS structured dialogue peer support groups
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/124
Other Adverse Events (participants affected / at risk) | 0/117 | 0/124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT04254198/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT04254198/SAP_001.pdf
  • Informed Consent Form (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT04254198/ICF_002.pdf